CLINICAL TRIAL: NCT06931717
Title: A Randomised Phase III Trial of Adjuvant Cemiplimab in Patients With Resected Stage II-IIIA NSCLC Who Have Not Received Prior Adjuvant Chemotherapy
Brief Title: A Clinical Study to Assess the Efficacy of Adjuvant Immunotherapy With Cemiplimab in Patients With Surgically Removed Non-small Cell Lung Cancer Who Have Not Received Prior Chemotherapy
Acronym: ARCH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 27-23
Record Dates: First submitted 2025-04-02; First posted 2025-04-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Stage II-IIIA NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Cemiplimab (Experimental): Cemiplimab, 350 mg i.v., every 3 weeks (±3 days), for 4 cycles, followed by 700 mg i.v., every 6 weeks (±1 week) for 6 cycles or until relapse or unacceptable toxicities, whichever occurs first.
  Interventions: Drug: Cemiplimab
- Control Arm: Observation (No Intervention): Observation.

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab, 350 mg i.v., every 3 weeks (±3 days), for 4 cycles, followed by 700 mg i.v., every 6 weeks (±1 week) for 6 cycles or until relapse or unacceptable toxicities, whichever occurs first.
  Arms: Experimental Arm: Cemiplimab

SUMMARY:
ARCH is a randomised, stratified, multicentre, phase III trial. Protocol treatment consists of cemiplimab, 350 mg i.v., every 3 weeks, for 4 cycles, followed by 700 mg i.v., every 6 weeks for 6 cycles or until relapse or unacceptable toxicities, whichever occurs first. The primary objective of the study is to determine the efficacy of adjuvant cemiplimab, as measured by disease-free survival, in patients without prior adjuvant platinum-based chemotherapy, compared to observation without adjuvant treatment. The primary objective will be assessed in patients with tumours with centrally confirmed PD-L1 expression of ≥1%.

ELIGIBILITY:
Inclusion Criteria:

* Pathological stage II-IIIA (UICC/ AJCC staging 9th edition) NSCLC Brain imaging should have been performed to complete staging, either preoperatively or postoperatively. If brain imaging has not been performed, a contrast-enhanced CT or MRI of the brain must be performed at screening prior randomisation.
* Complete resection with negative surgical margins (R0).

  * Acceptable types of surgical resection include any of the following:
* Lobectomy, sleeve lobectomy, bilobectomy, or pneumectomy.
* Segmentectomy for tumours ≤2 cm is permitted in patients with poor pulmonary reserve or another major comorbidity that contraindicates lobectomy.

  * Wedge resection is not allowed.
  * Lymph node dissection should be done according to applicable guidelines.
  * No disease recurrence following surgical resection.
* Tumour PD-L1 expression of ≥1%, determined locally using a locally approved immuno-histochemistry test.
* Availability of archival FFPE tumour tissue for central PD-L1 expression testing.
* Patient is not considered for adjuvant platinum-based chemotherapy due to:

  * Documented patient refusal; or
  * Patient is unfit to receive adjuvant platinum-based chemotherapy (per investigator assessment) due to:

ECOG PS2, or ECOG PS 0/1 and aged ≥70 years with substantial comorbidities or other contraindication(s) to platinum-based doublet chemotherapy.

* Estimated life expectancy of ≥3 months.
* Age ≥18 years.
* Patient has recovered from surgery-related complications.
* Adequate haematological, renal and liver function.
* Patient is able to comply with the trial protocol, in the investigator's judgment.
* Negative pregnancy test Female participants of childbearing potential (including women who had their last menstruation in the last 2 years), must have a negative serum pregnancy test within 5 weeks before randomisation. Pregnancy test must be repeated within 3 days before the first dose of protocol treatment and at every treatment visit (urine beta HCG test is sufficient).
* Use of highly effective contraceptive methods Female participants of childbearing potential (including women who had their last menstruation in the last 2 years) and male participants with a female partners of childbearing potential must agree to use a highly effective method of contraception for the duration of the protocol treatment and until 4 months after the last dose of cemiplimab.
* Written Informed Consent must be signed and dated by the patient and the investigator prior to any trial-related intervention.

Exclusion Criteria:

* EGFR-mutant or ALK-rearranged NSCLC.
* Any small cell component
* Prior neoadjuvant and/or adjuvant systemic treatment for NSCLC.

Note: Previous treatment for another malignancy not excluded as per next criterion (Participating in another interventional clinical trial for NSCLC) is allowed if the below conditions are fulfilled:

* Treatment with an approved systemic therapy is completed >4 weeks before randomisation or
* Treatment with systemic biologic therapy is completed >5 half-lives before randomisation and patient has recovered from any immune-mediated adverse events and endocrinopathies are adequately managed with hormone replacement.

  * Participating in another interventional clinical trial for NSCLC.
  * Diagnosis with another malignancy other than NSCLC that is progressing or requires active treatment.

Exceptions:

* Non-melanoma skin cancer that has undergone potentially curative therapy
* In situ cervical carcinoma
* Any tumour that has been deemed to be definitively treated, such as definitively treated non-metastatic prostate cancer.

  * Has any condition requiring ongoing/continuous corticosteroid therapy (>10 mg prednisone/day or anti-inflammatory equivalent) within 1 week prior to randomisation. Physiologic replacement doses are allowed even if they are >10 mg of prednisone per day or equivalent, as long as they are not being administered for immunosuppressive intent. Inhaled or topical steroids are permitted, provided that they are not for treatment of an autoimmune disorder.

Note: Patients who require a brief course of steroids (ex. 3 days in the week before randomisation) or physiologic replacement are allowed to be included in the study.

* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments.

The following are not exclusions: vitiligo, childhood asthma that has resolved, endocrinopathies (such as hypothyroidism or type 1 diabetes) that require only hormone replacement, or psoriasis that does not require systemic treatment.

* Encephalitis, meningitis, organic brain disease (e.g., Parkinson's disease) or uncontrolled seizures within 1 year prior to randomisation.
* Myocardial infarction within 6 months prior to randomisation.
* Known history of, or any evidence of, interstitial lung disease or active, non-infectious pneumonitis within 5 years prior to randomisation.
* Uncontrolled infection with HIV, hepatitis B, or hepatitis C infection; or the patient has a diagnosis of immunodeficiency.

  * Patients with known HIV infection who have controlled infection [undetectable viral load (HIV RNA PCR) and CD4 count above 350 either spontaneously or on a stable antiviral regimen] are allowed to be included in the study. Patients with controlled HIV infection should be monitored according to local standards.
  * Patients with hepatitis B (HBsAg+) with controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection and receiving antiviral therapy for hepatitis B) may be included in the study. Patients with controlled infection must undergo regular monitoring of HBV DNA. Patients must remain on antiviral therapy for at least 6 months after the last dose of cemiplimab.
  * Patients who are hepatitis C virus antibody positive (HCV Ab+) with controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) may be included in the study.
* Any infection requiring hospitalisation or treatment with intravenous anti-infectives within 2 weeks before randomisation.
* Receipt of a live vaccine within 28 days before randomisation.
* Receipt of a COVID-19 vaccination within 1 week before randomisation.
* Prior allogeneic stem cell transplantation or received organ transplants at any time, or autologous stem cell transplantation within 12 weeks before randomisation.
* Known or suspected hypersensitivity to cemiplimab or its excipients.
* Women who are pregnant, planning to become pregnant or are in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.
* Patients who are, or have an immediate family member who is, a member of the clinical study team, unless prior approval has been obtained from the sponsor (ETOP IBCSG Partners Foundation).
* Judgement by the investigator that the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From the date of randomisation until disease recurrence (including loco-regional recurrence, a distant (metastatic) recurrence or a second primary) or death from any cause. Assessed for approximately up to 59 months.
  Disease free survival (in patients with tumours with centrally confirmed PD-L1 expression of ≥1%).

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomisation until death from any cause. Assessed for approximately up to 59 months.
  OS is defined as the time from the date of randomisation until death from any cause. Censoring (for patients who are not reported as having died) will occur at the date last known to be alive. Patients without post-randomisation information will be censored at the date of randomisation (plus 1 day).
Incidence, nature and severity of adverse events according to CTCAE v5. | From the date the patient has signed the Informed Consent until the trial end. Assessed for approximately up to 59 months.
  All safety parameters will be summarised in tables to evaluate the toxicity/safety profile of the protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Soo, MB BS, PhD, FRACP, Study Chair — National University Hospital, Singapore; Patrick Forde, MD, MBBCh, PhD, Study Chair — Trinity St James Cancer Institute, Dublin, Ireland; Servet Bölükbas, MHBA, FETCS, FEBTS, FCCP, Study Chair — Universitätsmedizin Essen - Ruhrlandklinik Lungenkrebszentrum am Westdeutsches Tumorzentrum (LWTZ), Essen, Germany
Locations (34):
- Wien AKH, Vienna, Austria
- North Estonia Medical Centre Foundation, Talinn, Estonia
- France (2):
  - CHU d'Angers, Angers
  - Centre hospitalier d'Avignon, Avignon
- Germany (4):
  - Evangelische Lungenklinik Berlin, Buch
  - Ruhrlandklinik Essen, Essen
  - LMU München, München
  - Pius Hospital, University Medicine Oldenburg, Oldenburg
- Ireland (2):
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
- Italy (11):
  - SS Antonio e Biagio e Cesare Arrigo Hospital, Alessandria
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Instituto Europeo di Oncologia (IEO), Milan
  - AOU Maggiore della Carità, Novara
  - Instituto Oncologico Veneto IRCCS, Padua
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - University of Perugia, AO SM Misericorida Perugia, Perugia
  - Azienda ospedaliero-universitaria Senese Siena, Siena
  - AULSS2 Marca Trevigiana Treviso, Treviso
  - Universita di Verona - Department of Medicine, Verona
- National University Hospital, Singapore, Singapore
- Spain (10):
  - Complejo Hospitalario Universitario, A Coruña
  - Hospital General Universitario Dr. Balmis de Alicante, Alicante
  - Hospital Universitario Cruces, Barakaldo
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Clínico San Cecilio de Granada, Granada
  - Hospital Universitario de Jerez de La Frontera, Jerez de la Frontera
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital General Universitario de Valencia, Valencia
- Switzerland (2):
  - University Hospital Basel, Basel
  - Kantonsspital Winterthur, Winterthur